CLINICAL TRIAL: NCT04405323
Title: Interventional, Open-label, Randomized, Two-sequence Study Evaluating the Effect of CYP3A4 Inhibition on the Pharmacokinetics, Safety and Tolerability of Lu AG06466 in Healthy Men and Women
Brief Title: Study That Evaluates the Effect of CYP3A4 Inhibition on Lu AG06466 in Healthy Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18453A
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lu AG06466 - Sequence 1 (Experimental): Dosing on Days 1 and 8 will be following an overnight fast, and dosing on Days 3 and 10 will be following a standard high-fat breakfast.
  Interventions: Drug: Lu AG06466; Drug: Itraconazole
- Lu AG06466 - Sequence 2 (Experimental): Dosing on Days 1 and 8 will be following, a standard high-fat breakfast and dosing on Days 3 and 10 will be following an overnight fast.
  Interventions: Drug: Lu AG06466; Drug: Itraconazole

INTERVENTIONS:
Drug: Lu AG06466 — hard capsules, orally, single doses
Drug: Itraconazole — 200 and 300 mg, capsules, orally

SUMMARY:
A study to learn how a drug (itraconazole) that is known to inhibit a certain enzym in the liver, impacts the body's ability to breakdown Lu AG06466 into breakdown products in healthy men and women. The main breakdown product is Lu AG06988.

DETAILED DESCRIPTION:
Two sequence study where Lu AG06466 will be dosed with and without food, Sequence 1 and Sequence 2. Each subject will receive single oral doses of Lu AG06466. Subject will be randomized to one of two sequences.

For inhibition of CYP3A4, each subject will receive a once daily dosage of itraconazole from Day 5 to Day 11.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a BMI ≥18.5 and ≤30 kg/m2
* The subject is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, a neurological examination, vital signs, an electrocardiogram (ECG), and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.
* The subject must not be of childbearing potential (if a woman) or should use contraception (both sexes). If women, the subject must not be pregnant or breastfeeding.

Exclusion Criteria:

* The subject is a poor metabolizer (PM) of CYP2C9 and/or CYP2C19.

Other in- and exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
AUC(0-inf) Lu AG06466 | From 0 to 48 hours post-dose on Day 1, 3, 8 and 10
  Area under the Lu AG06466 plasma concentration-time curve from time zero to infinity
AUC(0-inf) Lu AG06988 | From 0 to 48 hours post-dose on Day 1, 3, 8 and 10
  Area under the Lu AG06988 plasma concentration-time curve from time zero to infinity
Cmax Lu AG06466 | From 0 to 48 hours post-dose on Day 1, 3, 8 and 10
  Maximum observed plasma concentration (Cmax) of Lu AG06466
Cmax Lu AG06988 | From 0 to 48 hours post-dose on Day 1, 3, 8 and 10
  Maximum observed plasma concentration (Cmax) of Lu AG06988

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- US1517, Miami, Florida, United States